CLINICAL TRIAL: NCT02828592
Title: A Study of T-Cell Replete, HLA-Mismatched Haploidentical Bone Marrow Transplantation With Post-Transplant Cyclophosphamide for Patients With Severe Aplastic Anemia Lacking HLA-Matched Related Donor
Brief Title: Haploidentical Bone Marrow Transplant With Post-Transplant Cyclophosphamide for Patients With Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1158
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Severe Aplastic Anemia
Keywords: SAA
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine; Cyclophosphamide; Whole-Body Irradiation; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flu/Cy/TBI (Experimental): Fludarabine, Cyclophosphamide, TBI followed by bone marrow transplantation. Post-transplant Cyclophosphamide will be on Days 3 & 4.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: Rabbit ATG

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2 IV QD x 5 days (Days -6 to -2)
Drug: Cyclophosphamide — 14.5 mg/kg/day IV x 2 doses (Days -6 & -5)
Radiation: Total Body Irradiation — 300 cGy x1 dose (Day -1)
  Other Names: TBI
Drug: Rabbit ATG — 1.5 mg/kg/day x 3 days (Days -3 to -1)
Drug: Cyclophosphamide — Post-transplant: 50 mg/kg IV QD (Day +3 to +4)

SUMMARY:
Severe aplastic anemia is a rare and serious form of bone marrow failure related to an immune-mediated mechanism that results in severe pancytopenia and high risk for infections and bleeding. Patients with matched sibling donors for transplantation have a 80-90% chance of survival; however, a response rate with just immunosuppression for those patients lacking suitable HLA-matched related siblings is only 60%. With immunosuppression, only 1/3 of patients are cured, 1/3 are dependent on long term immunosuppression, and the other 1/3 relapse or develop a clonal disorder. Recent studies have shown that using a haploidentical donor for transplantation has good response rates and significantly lower rates of acute and chronic GVHD.

DETAILED DESCRIPTION:
Mismatched haploidentical donors will be identified for patients with severe aplastic anemia. These patients will undergo a preparative regimen of Fludarabine/Cyclophosphamide/TBI followed by haploidentical bone marrow transplantation. Post-transplant Cyclophosphamide will be administered on Days 3 & 4. Immunosuppression with Tacrolimus and MMF will begin on Day +5; MMF will be discontinued on Day +35 while Tacrolimus continues until Day +180. Investigators hypothesize that haploidentical transplantation with the above-mentioned preparative regimen will have a <30% graft failure rate. The one-sided exact Binomial test at 5% significance level will be used to test this hypothesis. The size of 20 patients provides the power of 92.5% for confirming the 30-day graft failure rate <30%.

ELIGIBILITY:
Inclusion Criteria:

* Availability of 3/6 - 5/6 matched (HLA-A, B, DR) related donor who must have negative HLA cross-match in the host vs. graft direction
* Age <= 65 years for previously treated and <= 75 years for previously treated patients
* KPS >= 70%
* Aplastic Anemia that meets the following criteria:

Peripheral Blood (must fulfill 2 of 3):

* <500 PMN/mm3
* <20,000 platelets
* absolute reticulocyte count <40,000/microL

Bone Marrow (must be either):

* markedly hypocellular (<25% of normal cellularity)
* moderately hypocellular with 70% non-myeloid precursors and patient meets peripheral blood criteria above

Exclusion Criteria:

* poor cardiac function (LVEF <40%)
* poor pulmonary function (FEV1 & FVC <50% predicted)
* poor liver function (bili >= 2mg/dL)
* poor renal function (creatinine >= 2.0mg/dL or creatinine clearance <40mL/min)
* prior allogeneic transplant

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrate sustained engraftment after T-cell replete HLA-mismatched haploidentical bone marrow transplantation by collecting chimerism tests monthly following transplant | 2 years
  Hypothesis is that following preparative regimen and bone marrow transplantation, the 30-day graft failure rate will be <30%.

SECONDARY OUTCOMES:
Determine the incidence of regimen-related mortality at 100 days post transplantation by recording treatment-related adverse events | 2 years
Determine the incidence of grade 2-4 and 3-4 acute graft versus host disease at 100 days post transplantation by assessing signs and symptoms of GVHD throughout post-transplant course | 2 years
Determine incidence of chronic GVHD at 6 months and 1 year post transplantation by assessing signs and symptoms of GVHD throughout post-transplant course | 2 years
Estimate overall survival at 100 days and 1 year post transplantation by collecting survival information at those time points | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Melhem Solh, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (2):
- United States (2):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brodsky RA, Chen AR, Dorr D, Fuchs EJ, Huff CA, Luznik L, Smith BD, Matsui WH, Goodman SN, Ambinder RF, Jones RJ. High-dose cyclophosphamide for severe aplastic anemia: long-term follow-up. Blood. 2010 Mar 18;115(11):2136-41. doi: 10.1182/blood-2009-06-225375. Epub 2009 Dec 16. PMID 20018919
- [Result] Socie G. Allogeneic BM transplantation for the treatment of aplastic anemia: current results and expanding donor possibilities. Hematology Am Soc Hematol Educ Program. 2013;2013:82-6. doi: 10.1182/asheducation-2013.1.82. PMID 24319167
- [Result] Young NS. Current concepts in the pathophysiology and treatment of aplastic anemia. Hematology Am Soc Hematol Educ Program. 2013;2013(1):76-81. doi: 10.1182/asheducation-2013.1.76. PMID 24319166
- [Result] Scheinberg P, Young NS. How I treat acquired aplastic anemia. Blood. 2012 Aug 9;120(6):1185-96. doi: 10.1182/blood-2011-12-274019. Epub 2012 Apr 19. PMID 22517900
- [Result] Bashey A, Zhang X, Jackson K, Brown S, Ridgeway M, Solh M, Morris LE, Holland HK, Solomon SR. Comparison of Outcomes of Hematopoietic Cell Transplants from T-Replete Haploidentical Donors Using Post-Transplantation Cyclophosphamide with 10 of 10 HLA-A, -B, -C, -DRB1, and -DQB1 Allele-Matched Unrelated Donors and HLA-Identical Sibling Donors: A Multivariable Analysis Including Disease Risk Index. Biol Blood Marrow Transplant. 2016 Jan;22(1):125-33. doi: 10.1016/j.bbmt.2015.09.002. Epub 2015 Sep 7. PMID 26359881
- [Result] Solomon SR, Sizemore CA, Sanacore M, Zhang X, Brown S, Holland HK, Morris LE, Bashey A. Total Body Irradiation-Based Myeloablative Haploidentical Stem Cell Transplantation Is a Safe and Effective Alternative to Unrelated Donor Transplantation in Patients Without Matched Sibling Donors. Biol Blood Marrow Transplant. 2015 Jul;21(7):1299-307. doi: 10.1016/j.bbmt.2015.03.003. Epub 2015 Mar 19. PMID 25797174
- [Result] Bashey A, Solomon SR. T-cell replete haploidentical donor transplantation using post-transplant CY: an emerging standard-of-care option for patients who lack an HLA-identical sibling donor. Bone Marrow Transplant. 2014 Aug;49(8):999-1008. doi: 10.1038/bmt.2014.62. Epub 2014 May 19. PMID 24842530
- [Result] Rozman C, Marin P, Nomdedeu B, Montserrat E. Criteria for severe aplastic anaemia. Lancet. 1987 Oct 24;2(8565):955-7. doi: 10.1016/s0140-6736(87)91432-2. PMID 2889870
- [Result] Atta EH, de Sousa AM, Schirmer MR, Bouzas LF, Nucci M, Abdelhay E. Different outcomes between cyclophosphamide plus horse or rabbit antithymocyte globulin for HLA-identical sibling bone marrow transplant in severe aplastic anemia. Biol Blood Marrow Transplant. 2012 Dec;18(12):1876-82. doi: 10.1016/j.bbmt.2012.07.004. Epub 2012 Jul 11. PMID 22796534